CLINICAL TRIAL: NCT02638337
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Multicenter Study to Evaluate the Efficacy and Safety of Ospemifene in Patients With Moderate to Severe Vaginal Dryness, a Symptom of Vulvo-vaginal Atrophy (VVA) Due to Menopause
Brief Title: Study to Evaluate Ospemifene in Patients With Moderate to Severe Vaginal Dryness Due to Menopause
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1517I0231
Record Dates: First submitted 2015-12-18; First posted 2015-12-23 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Vaginal Dryness
Keywords: Vulvo-vaginal Atrophy; menopause
MeSH Terms: interventions — Ospemifene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ospemifene (Experimental): Participants will take one tablet of ospemifene 60 mg orally, once a day for 12 weeks.
  Interventions: Drug: Ospemifene
- Placebo (Placebo Comparator): Participants will take one tablet of matching placebo, orally, once a day for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ospemifene — 60 mg tablet
  Other Names: Osphena®
  Arms: Ospemifene
Drug: Placebo — Tablet identical to the ospemifene tablet without drug
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of ospemifene 60 mg once daily (QD) compared with placebo in treatment of vulvo-vaginal atrophy (VVA) due to menopause in women with moderate to severe vaginal dryness as the most bothersome symptom (MBS) of VVA.

ELIGIBILITY:
Inclusion Criteria:

* Subject is postmenopausal.
* Subject has moderate to severe vaginal dryness as the self-reported MBS of VVA.

Exclusion Criteria:

* Subject has clinically significant abnormal findings in the physical examination.
* Subject has a body mass index (BMI) equal to or greater than 38 kg/m^2
* Subject has uncontrolled hypertension.
* Subject has clinically significant abnormal findings in the gynecological examination other than signs of vaginal atrophy.
* Subject has uterine/vaginal bleeding of unknown origin.
* Subject has a vaginal infection requiring medication (may be treated and be eligible for study).

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi

REFERENCES:
- [Derived] Lara LA, Cartagena-Ramos D, Figueiredo JB, Rosa-E-Silva ACJ, Ferriani RA, Martins WP, Fuentealba-Torres M. Hormone therapy for sexual function in perimenopausal and postmenopausal women. Cochrane Database Syst Rev. 2023 Aug 24;8(8):CD009672. doi: 10.1002/14651858.CD009672.pub3. PMID 37619252
- [Derived] Archer DF, Goldstein SR, Simon JA, Waldbaum AS, Sussman SA, Altomare C, Zhu J, Yoshida Y, Schaffer S, Soulban G. Efficacy and safety of ospemifene in postmenopausal women with moderate-to-severe vaginal dryness: a phase 3, randomized, double-blind, placebo-controlled, multicenter trial. Menopause. 2019 Jan 28;26(6):611-621. doi: 10.1097/GME.0000000000001292. PMID 30694917

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized at 68 sites in the United States.
Pre-assignment Details: After a screening period of up to 4 weeks, participants who met all eligibility criteria were randomized in a 1:1 ratio to receive either ospemifene 60 mg once daily or matching placebo for 12 weeks. Randomization was stratified by severity of most bothersome symptom of vaginal dryness on Day 1 and by the presence or absence of the uterus.
Groups:
- Ospemifene: Participants received one tablet of ospemifene 60 mg orally, once a day for 12 weeks.
- Placebo: Participants received one tablet of matching placebo, orally, once a day for 12 weeks.
Period: Overall Study
Arm/Group | Ospemifene | Placebo
Started | 316 | 315
Received Treatment | 313 | 315
Completed | 283 | 279
Not Completed | 33 | 36
Not completed — Adverse Event | 6 | 10
Not completed — Protocol Violation | 3 | 0
Not completed — Withdrawal by Subject | 13 | 16
Not completed — Lost to Follow-up | 7 | 7
Not completed — Other - Miscellaneous | 4 | 3

BASELINE CHARACTERISTICS:
Population: The intent-to-treat population included participants who received at least 1 dose of study drug. One participant who enrolled at 2 different sites was excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ospemifene | Placebo | Total
Number analyzed (Participants) | 313 | 314 | 627
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (6.6) | 59.8 (7.2) | 59.7 (6.9)
Age, Customized [Count of Participants; unit: Participants]
  >= 40 to < 45 years | 3 | 7 | 10
  >= 45 to < 55 years | 66 | 58 | 124
  >= 55 to < 65 years | 171 | 174 | 345
  >= 65 years | 73 | 75 | 148
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 313 | 314 | 627
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 84 | 79 | 163
  Not Hispanic or Latino | 228 | 234 | 462
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 7 | 7
  Asian | 1 | 3 | 4
  Black or African American | 38 | 32 | 70
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 273 | 266 | 539
  Other | 1 | 6 | 7
Presence of Uterus [Count of Participants; unit: Participants]
  Yes | 128 | 132 | 260
  No | 185 | 182 | 367
Current Hot Flashes [Count of Participants; unit: Participants]
  Yes | 26 | 28 | 54
  No | 287 | 286 | 573
Previous Hormone Treatment as Prior Treatment [Count of Participants; unit: Participants]
  None | 305 | 307 | 612
  Oral | 5 | 5 | 10
  Transdermal | 0 | 0 | 0
  Vaginal | 4 | 3 | 7
  Other | 0 | 0 | 0
Duration of Vulvovaginal Atrophy (VVA) [Mean (Standard Deviation); unit: years] | 8.36 (6.92) | 8.98 (7.79) | 8.67 (7.37)
Percentage of Parabasal Cells in the Vaginal Squamous Epithelium: [Mean (Standard Deviation); unit: percentage of cells] — The percentage of each of the 3 main types of vaginal epithelial cells (parabasal, intermediate, and superficial) indicates the degree of maturation attained by the vaginal epithelium and can be used to detect hormonal effects in menopausal and postmenopausal women. Parabasal cells are immature squamous cells in the lining of the vagina. A predominance of parabasal cells indicates absence of estrogenic stimulation.
  Vaginal smear samples were taken from the middle third of the lateral vaginal wall and were evaluated at a central laboratory by a qualified pathologist. Population: Participants in the intent-to-treat population with available data
  percentage of cells
    number analyzed (Participants) | 306 | 308 | 614
    (all) | 25.8 (33.3) | 28.3 (33.1) | 27.0 (33.2)
Percentage of Superficial Cells in the Vaginal Squamous Epithelium [Mean (Standard Deviation); unit: percentage of cells] — The percentage of each of the 3 main types of vaginal epithelial cells (parabasal, intermediate, and superficial) indicates the degree of maturation attained by the vaginal epithelium and can be used to detect hormonal effects in menopausal and postmenopausal women. Superficial cells are mature squamous cells in the lining of the vagina; a predominance of superficial cells indicates the presence of estrogen.
  Vaginal smear samples were taken from the middle third of the lateral vaginal wall and were evaluated at a central laboratory by a qualified pathologist. Population: Participants in the intent-to-treat population with available data
  percentage of cells
    number analyzed (Participants) | 306 | 308 | 614
    (all) | 3.0 (7.6) | 2.8 (6.9) | 2.9 (7.2)
Vaginal pH [Mean (Standard Deviation); unit: pH] — A typical vaginal pH in women of reproductive age is between 3.5 and 4.5, increasing to > 4.5 after menopause.
  pH | 6.11 (0.70) | 6.14 (0.73) | 6.12 (0.71)
Mean Severity of Most Bothersome Symptom of Vaginal Dryness [Mean (Standard Deviation); unit: units on a scale] — The severity of the most bothersome symptom of vaginal dryness was assessed by the participant through the VVA questionnaire as none = 0, mild = 1, moderate = 2, and severe = 3.
  units on a scale | 2.53 (0.50) | 2.54 (0.50) | 2.54 (0.5)
Severity of Most Bothersome Symptom of Vaginal Dryness [Count of Participants; unit: Participants] — The severity of the most bothersome symptom of vaginal dryness was assessed by the participant through the VVA questionnaire as none = 0, mild = 1, moderate = 2, and severe = 3.
  Participants
    None | 0 | 0 | 0
    Mild | 0 | 0 | 0
    Moderate | 148 | 143 | 291
    Severe | 165 | 171 | 336

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Percentage of Parabasal Cells in the Maturation Index of the Vaginal Smear at Week 12
Description: Parabasal cells are immature squamous cells in the lining of the vagina. A predominance of parabasal cells indicates absence of estrogenic stimulation and vaginal atrophy.
  Vaginal smear samples were taken from the middle third of the lateral vaginal wall and were evaluated at a central laboratory by a qualified pathologist.
  A decrease in parabasal cells indicates improvement in vaginal atrophy. To calculate least squares (LS) means, a mixed-effects model for repeated measures (MMRM) model was used.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available baseline data
Measure: Least Squares Mean (Standard Error); unit: percentage of cells
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 306 | 308
percentage of cells | -23.7 (1.4) | -1.9 (1.4)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; For the percentage of parabasal cells a mixed-effects model for repeated measures (MMRM) approach was used, with repeated measurements of the change from baseline as the response variable; treatment, week, treatment by week interaction, and study center as fixed effects; and baseline value modeled as a covariate; Test type: Superiority; p < 0.0001, Mixed-effects model repeated measures; MMRM model with treatment, week, treatment by week interaction, and study center as fixed effects; and baseline value modeled as a covariate; LS Mean Difference = -21.8, 95% CI 2-sided [-25.7 to -18.0]

2. Primary Outcome: Change From Baseline in the Percentage of Superficial Cells in the Maturation Index of the Vaginal Smear at Week 12
Description: Superficial cells are mature squamous cells in the lining of the vagina that can decrease in number after menopause resulting in vulvovaginal atrophy.
  Vaginal smear samples were taken from the middle third of the lateral vaginal wall and were evaluated at a central laboratory by a qualified pathologist.
  An increase in the number of superficial cells indicates improvement in atrophy.
  To calculate least squares (LS) means, a mixed-effects model for repeated measures (MMRM) model was used.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available baseline data
Measure: Least Squares Mean (Standard Error); unit: percentage of cells
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 306 | 308
percentage of cells | 7.8 (0.7) | 0.6 (0.7)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Test type: Superiority; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 7.2, 95% CI 2-sided [5.2 to 9.1]

3. Primary Outcome: Change From Baseline in the Vaginal pH at Week 12
Description: The pH scale ranges from 0 to 14. A pH of 7 is neutral, less than 7 is acidic, and greater than 7 is basic. A typical vaginal pH in women of reproductive age is between 3.5 and 4.5, increasing to > 4.5 after menopause.
  Vaginal pH was measured by the investigator using a pH indicator strip at the middle third of the vaginal wall.
  To calculate least squares (LS) means, a mixed-effects model for repeated measures (MMRM) model was used.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available baseline data
Measure: Least Squares Mean (Standard Error); unit: pH
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 313 | 314
pH | -1.01 (0.04) | -0.29 (0.04)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Test type: Superiority; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.72, 95% CI 2-sided [-0.84 to -0.59]

4. Primary Outcome: Change From Baseline in the Severity of Self-reported Most Bothersome Symptom (MBS) of Vaginal Dryness at Week 12
Description: The severity of the most bothersome symptom of vaginal dryness was assessed by the participant through the VVA questionnaire as none = 0, mild = 1, moderate = 2, and severe = 3.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available baseline data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 313 | 314
units on a scale | -1.29 (1.01) | -0.91 (0.96)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; For the MBS of vaginal dryness a generalized estimating equations (GEE) model was used to fit a marginal proportional odds model to the longitudinal ordered categorical data, with repeated measurements of the change from baseline as the response variable; treatment, week, treatment by week interaction, and study center as fixed effects; and baseline severity of dryness modeled as a covariate; Test type: Superiority; p < 0.0001, Generalized estimating equations model; GEE model with treatment, week, treatment by week interaction, and study center as fixed effects and baseline severity of dryness as a covariate; Odds Ratio (OR) = 2.23, 95% CI 2-sided [1.62 to 3.06] — Odds ratio is the exponential of the mean of cumulative log odds ratio

5. Primary Outcome: Number of Participants With Adverse Events
Description: Treatment-related adverse events (AEs) were defined as AEs that were considered by the investigator to be related to investigational medicinal product, for which causal relationship with the study drug could be reasonably explained.
  A serious adverse event (SAE) is defined as any AE occurring at any dose that resulted in any of the following outcomes:
  * Death
  * Life-threatening condition
  * Hospitalization or prolongation of existing hospitalization for treatment
  * Persistent or significant disability/incapacity
  * Congenital anomaly/birth defect
  * Other medically important conditions that, based on medical judgment, may jeopardize the participant's health and may require medical intervention to prevent one of the outcomes listed above.
Time Frame: From the first dose of study drug up to 14 days after the last dose; 14 weeks
Population: Participants who received at least 1 dose of study drug. Four participants randomized to placebo received ospemifene in error and are counted in the ospemifene group for safety assessments. One participant randomized to placebo who enrolled at 2 different sites at the same time was excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 317 | 310
Participants
  Any adverse event | 112 | 103
  Treatment-related adverse events | 28 | 20
  Adverse events leading to withdrawal | 6 | 10
  Treatment-related AEs leading to withdrawal | 5 | 3
  Serious adverse events | 5 | 3
  Treatment-related serious adverse events | 0 | 0
  Adverse events with outcome of death | 0 | 0

6. Secondary Outcome: Change From Baseline in the Percentage of Parabasal Cells in the Maturation Index of the Vaginal Smear at Weeks 4 and 8
Description: Parabasal cells are immature squamous cells in the lining of the vagina. A predominance of parabasal cells indicates absence of estrogenic stimulation and vaginal atrophy. Vaginal smear samples were taken from the middle third of the lateral vaginal wall and were evaluated at a central laboratory by a qualified pathologist. A decrease in parabasal cells indicates improvement in vaginal atrophy.
Time Frame: Baseline and Weeks 4 and 8
Population: Intent-to-treat population with baseline data
Measure: Least Squares Mean (Standard Error); unit: percentage of cells
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 306 | 308
percentage of cells
  Week 4 | -21.6 (1.3) | 0.0 (1.3)
  Week 8 | -23.7 (1.3) | -1.9 (1.3)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Week 4; Test type: Superiority; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -21.6, 95% CI 2-sided [-25.2 to -18.0]
Statistical Analysis 2: Comparison: Ospemifene vs Placebo; Week 8; Test type: Superiority; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -21.8, 95% CI 2-sided [-25.4 to -18.1]

7. Secondary Outcome: Change From Baseline in the Percentage of Superficial Cells in the Maturation Index of the Vaginal Smear at Weeks 4 and 8
Description: Superficial cells are mature squamous cells in the lining of the vagina that can decrease in number after menopause resulting in vulvovaginal atrophy. Vaginal smear samples were taken from the middle third of the lateral vaginal wall and were evaluated at a central laboratory by a qualified pathologist. An increase in the number of superficial cells indicates improvement in atrophy.
Time Frame: Baseline and Weeks 4 and 8
Population: Intent-to-treat population with available baseline data
Measure: Least Squares Mean (Standard Error); unit: percentage of cells
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 306 | 308
percentage of cells
  Week 4 | 5.6 (0.6) | -0.2 (0.6)
  Week 8 | 7.1 (0.7) | -0.2 (0.6)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Week 4; Test type: Superiority; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 5.8, 95% CI 2-sided [4.2 to 7.3]
Statistical Analysis 2: Comparison: Ospemifene vs Placebo; Week 8; Test type: Superiority; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = 7.2, 95% CI 2-sided [5.5 to 9.0]

8. Secondary Outcome: Change From Baseline in the Vaginal pH
Description: The pH scale ranges from 0 to 14. A pH of 7 is neutral, less than 7 is acidic, and greater than 7 is basic. A typical vaginal pH in women of reproductive age is between 3.5 and 4.5, increasing to > 4.5 after menopause. Vaginal pH was measured by the investigator using a pH indicator strip at the middle third of the vaginal wall.
Time Frame: Baseline and Weeks 4 and 8
Population: Intent-to-treat population with available baseline data
Measure: Least Squares Mean (Standard Error); unit: pH
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 313 | 314
pH
  Week 4 | -0.81 (0.04) | -0.24 (0.04)
  Week 8 | -0.95 (0.04) | -0.32 (0.04)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Week 4; Test type: Superiority; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.58, 95% CI 2-sided [-0.69 to -0.46]
Statistical Analysis 2: Comparison: Ospemifene vs Placebo; Week 8; Test type: Superiority; p < 0.0001, Mixed-effects model repeated measures; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.63, 95% CI 2-sided [-0.75 to -0.51]

9. Secondary Outcome: Change From Baseline in the Severity of Self-reported Most Bothersome Symptom (MBS) of Vaginal Dryness at Weeks 4 and 8
Description: as for outcome 4
Time Frame: Baseline and Weeks 4 and 8
Population: Intent-to-treat population with available data at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 313 | 314
units on a scale
  Week 4 | -0.83 (0.90) | -0.62 (0.89)
  Week 8 | -1.14 (0.97) | -0.84 (0.95)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Week 4; Test type: Superiority; p = 0.0005, Generalized estimating equations model; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.27 to 2.36] — Odds ratio is the exponential of the mean of cumulative log odds ratio
Statistical Analysis 2: Comparison: Ospemifene vs Placebo; Week 8; Test type: Superiority; p < 0.0001, Generalized estimating equations model; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 2.01, 95% CI 2-sided [1.47 to 2.74] — Odds ratio is the exponential of the mean of cumulative log odds ratio

10. Secondary Outcome: Change From Baseline in Vaginal and/or Vulvar Irritation or Itching
Description: The severity of vaginal and/or vulvar irritation or itching was assessed by the participant through the VVA questionnaire as none = 0, mild = 1, moderate = 2, and severe = 3.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: Intent-to-treat population; participants whose baseline values were moderate or severe were included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 130 | 138
units on a scale
  Week 4 | -0.93 (1.00) | -0.99 (1.02)
  Week 8 | -1.17 (1.01) | -1.16 (1.04)
  Week 12 | -1.38 (1.00) | -1.40 (0.96)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Week 4; Test type: Superiority; p = 0.6263, Generalized estimating equations model; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.55 to 1.43] — Odds ratio is the exponential of the mean of cumulative log odds ratio
Statistical Analysis 2: Comparison: Ospemifene vs Placebo; Week 8; Test type: Superiority; p = 0.7869, Generalized estimating equations model; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.66 to 1.75] — Odds ratio is the exponential of the mean of cumulative log odds ratio
Statistical Analysis 3: Comparison: Ospemifene vs Placebo; Week 12; Test type: Superiority; p = 0.8894, Generalized estimating equations model; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.65 to 1.64] — Odds ratio is the exponential of the mean of cumulative log odds ratio

11. Secondary Outcome: Change From Baseline in Difficult or Painful Urination
Description: The severity of difficult or painful urination was assessed by the participant through the VVA questionnaire as none = 0, mild = 1, moderate = 2, and severe = 3.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: Intent-to-treat population; participants whose baseline values were moderate or severe were included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 40 | 37
units on a scale
  Week 4 | -1.23 (1.01) | -1.21 (0.84)
  Week 8 | -1.42 (0.95) | -1.15 (0.97)
  Week 12 | -1.56 (0.93) | -1.38 (0.91)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Week 4; Test type: Superiority; p = 0.8369, Generalized estimating equations model; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.40 to 2.10] — Odds ratio is the exponential of the mean of cumulative log odds ratio
Statistical Analysis 2: Comparison: Ospemifene vs Placebo; Week 8; Test type: Superiority; p = 0.3970, Generalized estimating equations model; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.58 to 3.95] — Odds ratio is the exponential of the mean of cumulative log odds ratio
Statistical Analysis 3: Comparison: Ospemifene vs Placebo; Week 12; Test type: Superiority; p = 0.5391, Generalized estimating equations model; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.54 to 3.26] — Odds ratio is the exponential of the mean of cumulative log odds ratio

12. Secondary Outcome: Change From Baseline in Vaginal Pain Associated With Sexual Activity
Description: The severity of vaginal pain associated with sexual activity was assessed by the participant through the VVA questionnaire as none = 0, mild = 1, moderate = 2, and severe = 3.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: Intent-to-treat population; participants whose baseline values were moderate or severe were included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 201 | 203
units on a scale
  Week 4 | -1.24 (1.11) | -0.99 (1.11)
  Week 8 | -1.41 (1.08) | -1.26 (1.13)
  Week 12 | -1.55 (1.05) | -1.21 (1.07)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Week 4; Test type: Superiority; p = 0.0095, Generalized estimating equations model; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.13 to 2.40] — Odds ratio is the exponential of the mean of cumulative log odds ratio
Statistical Analysis 2: Comparison: Ospemifene vs Placebo; Week 8; Test type: Superiority; p = 0.0542, Generalized estimating equations model; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.99 to 2.11] — Odds ratio is the exponential of the mean of cumulative log odds ratio
Statistical Analysis 3: Comparison: Ospemifene vs Placebo; Week 12; Test type: Superiority; p = 0.0004, Generalized estimating equations model; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.97, 95% CI 2-sided [1.35 to 2.88] — Odds ratio is the exponential of the mean of cumulative log odds ratio

13. Secondary Outcome: Change From Baseline in Vaginal Bleeding Associated With Sexual Activity
Description: The severity of vaginal bleeding associated with sexual activity was assessed by the participant through the VVA questionnaire as none = 0, mild = 1, moderate = 2, and severe = 3.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: Intent-to-treat population; participants whose baseline values were moderate or severe were included
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 51 | 37
units on a scale
  Week 4 | -1.17 (1.09) | -1.33 (1.14)
  Week 8 | -1.47 (0.92) | -1.58 (1.09)
  Week 12 | -1.55 (0.79) | -1.61 (1.06)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Week 4; Test type: Superiority; p = 0.4336, Generalized estimating equations model; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.30 to 1.67] — Odds ratio is the exponential of the mean of cumulative log odds ratio
Statistical Analysis 2: Comparison: Ospemifene vs Placebo; Week 8; Test type: Superiority; p = 0.7672, Generalized estimating equations model; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.37 to 2.08] — Odds ratio is the exponential of the mean of cumulative log odds ratio
Statistical Analysis 3: Comparison: Ospemifene vs Placebo; Week 12; Test type: Superiority; p = 0.7101, Generalized estimating equations model; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.39 to 1.89] — Odds ratio is the exponential of the mean of cumulative log odds ratio

14. Secondary Outcome: Change From Baseline in Maturation Value
Description: The maturation value is an indicator of the level of maturation attained by the vaginal epithelium.
  Vaginal smear samples were taken from the middle third of the lateral vaginal wall and were evaluated at the central laboratory by a qualified pathologist. Parabasal cells (P), intermediary cells (I), and superficial cells (S) were counted and results were expressed as the maturation value (MV), whereby superficial cells were assigned a point value of 1.0, intermediate cells were assigned a point value of 0.5, and parabasal cells were assigned a point value of 0. The maturation value (MV) was defined as:
  (percentage of superficial cells * 1) + (percentage of intermediate cells * 0.5) + (percentage of parabasal calls * 0).
  Lower MV indicates lower estrogen effect.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: Intent-to-treat population with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 306 | 308
units on a scale
  Week 4: number analyzed (Participants) | 241 | 266
  Week 4 | 13.33 (0.79) | -0.65 (0.75)
  Week 8: number analyzed (Participants) | 229 | 249
  Week 8 | 15.34 (0.82) | 0.61 (0.78)
  Week 12: number analyzed (Participants) | 216 | 233
  Week 12 | 16.19 (0.87) | 1.28 (0.83)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Week 4; Test type: Superiority; p < 0.0001, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = 13.98, 95% CI 2-sided [11.85 to 16.12]
Statistical Analysis 2: Comparison: Ospemifene vs Placebo; Week 8; Test type: Superiority; p < 0.0001, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = 14.73, 95% CI 2-sided [12.50 to 16.96]
Statistical Analysis 3: Comparison: Ospemifene vs Placebo; Week 12; Test type: Superiority; p < 0.0001, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = 14.91, 95% CI 2-sided [12.55 to 17.28]

15. Secondary Outcome: Percentage of Participants Who Were Responders at Week 4, Week 8, and Week 12
Description: A participant was defined as a responder if all the following conditions were met::
  * Increase from baseline in maturation value of at least 10
  * Decrease from baseline in vaginal pH of at least 0.5
  * Improvement from baseline (decrease in severity) of at least 1 point in the most bothersome symptom of vaginal dryness
Time Frame: Baseline and Weeks 4, 8, and 12
Population: Intent-to-treat population with available data at each time point
Measure: Number; unit: percentage of participants
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 313 | 314
percentage of participants
  Week 4: number analyzed (Participants) | 240 | 265
  Week 4 | 19.2 | 2.6
  Week 8: number analyzed (Participants) | 229 | 249
  Week 8 | 27.9 | 4.4
  Week 12: number analyzed (Participants) | 216 | 233
  Week 12 | 31.5 | 6.0
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Week 4; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 2: Comparison: Ospemifene vs Placebo; Week 8; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 3: Comparison: Ospemifene vs Placebo; Week 12; Test type: Superiority; p < 0.0001, Fisher Exact

16. Secondary Outcome: Change From Baseline in Vaginal Health Index
Description: The investigator performed an evaluation of the vagina, assessing overall elasticity, fluid secretion, pH, condition of epithelial mucosa, and moisture. The severity of each characteristic was assessed using a 5-grade scale from 1 (worst) to 5 (best). The total score was calculated as the sum of the 5 individual scores and ranges from 5 to 25, where higher scores indicate better vaginal health
Time Frame: Baseline and Weeks 4, 8, and 12
Population: Intent-to-treat population with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 312 | 312
units on a scale
  Week 4: number analyzed (Participants) | 297 | 295
  Week 4 | 3.9 (0.2) | 1.5 (0.2)
  Week 8: number analyzed (Participants) | 289 | 283
  Week 8 | 5.0 (0.2) | 2.1 (0.2)
  Week 12: number analyzed (Participants) | 277 | 278
  Week 12 | 5.2 (0.2) | 2.3 (0.2)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Week 4; Test type: Superiority; p < 0.0001, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = 2.5, 95% CI 2-sided [2.0 to 3.0]
Statistical Analysis 2: Comparison: Ospemifene vs Placebo; Week 8; Test type: Superiority; p < 0.0001, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = 2.9, 95% CI 2-sided [2.4 to 3.4]
Statistical Analysis 3: Comparison: Ospemifene vs Placebo; Week 12; Test type: Superiority; p < 0.0001, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = 2.8, 95% CI 2-sided [2.2 to 3.4]

17. Secondary Outcome: Change From Baseline in Vulvar Health Index
Description: The investigator performed a visual examination of the vulva, assessing the labia majora, labia minora, clitoris, introitus appearance and elasticity, color, discomfort and pain, and presence of other findings (eg, petechiae, excoriations, ulcers, etc). The severity of each characteristic was assessed on a 4-point scale as 0 = normal, 1 = mild, 2 = moderate, and 3 = severe. The total score was calculated by adding the 7 individual scores and ranges from 0 to 21, where lower scores indicate better vulvar health. A negative change from baseline indicates improvement.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: Intent-to-treat population with available data at each timepoint
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 308 | 308
units on a scale
  Week 4: number analyzed (Participants) | 290 | 287
  Week 4 | -2.2 (0.2) | -1.4 (0.2)
  Week 8: number analyzed (Participants) | 281 | 272
  Week 8 | -2.8 (0.2) | -1.7 (0.2)
  week 12: number analyzed (Participants) | 273 | 270
  week 12 | -2.8 (0.2) | -1.6 (0.2)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Week 4; Test type: Superiority; p = 0.0002, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = -0.8, 95% CI 2-sided [-1.3 to -0.4]
Statistical Analysis 2: Comparison: Ospemifene vs Placebo; Week 8; Test type: Superiority; p < 0.0001, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = -1.1, 95% CI 2-sided [-1.5 to -0.6]
Statistical Analysis 3: Comparison: Ospemifene vs Placebo; Week 12; Test type: Superiority; p < 0.0001, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = -1.2, 95% CI 2-sided [-1.6 to -0.7]

18. Secondary Outcome: Change From Baseline in Vulvovaginal Imaging Total Score at Week 12
Description: Vulvovaginal imaging was performed by trained site personnel following a standard procedure. Photographs were assessed by an Independent Panel Review (IPR) in a blinded fashion. Nine parameters (labia majora, labia minora, clitoris, urethra, introitus and elasticity, color, erythema, moisture, and other findings (petechiae, excoriation, ulceration, etc.)) were evaluated on a scale from 0 (normal/none) to 3 (severe). The total score was calculated from the sum of the 9 individual scores and ranged from 0 to 27 with lower values indicating better vulvovaginal health; a negative change from baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population; participants who agreed to participate in the optional vaginal imaging, and with available data at both time points were included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 135 | 141
units on a scale | -1.1 (0.3) | -0.1 (0.3)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Test type: Superiority; p = 0.0118, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = -1.0, 95% CI 2-sided [-1.8 to -0.2]

19. Secondary Outcome: Change From Baseline in Female Sexual Function Index Total Score
Description: The Female Sexual Function Index consists of 19 questions organized into 6 domains (desire, arousal, lubrication, orgasm, satisfaction, and pain) answered by the participant on a 5-point scale from 1 to 5. Where relevant, some questions also include an option of 0 if a question is not applicable due to no sexual activity. Each domain score was calculated by adding the scores of each item in the domain and multiplying by a domain factor. The total score was calculated by summing each domain score and ranges from 2 to 36, with higher values indicating better sexual function.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: Intent-to-treat population with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 303 | 308
units on a scale
  Week 4: number analyzed (Participants) | 285 | 286
  Week 4 | 4.13 (0.43) | 4.11 (0.43)
  Week 8: number analyzed (Participants) | 273 | 274
  Week 8 | 4.70 (0.49) | 4.51 (0.49)
  Week 12: number analyzed (Participants) | 261 | 271
  Week 12 | 5.71 (0.55) | 4.13 (0.54)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Week 4; Test type: Superiority; p = 0.9748, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = 0.02, 95% CI 2-sided [-1.17 to 1.20]
Statistical Analysis 2: Comparison: Ospemifene vs Placebo; Week 8; Test type: Superiority; p = 0.7865, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = 0.19, 95% CI 2-sided [-1.18 to 1.56]
Statistical Analysis 3: Comparison: Ospemifene vs Placebo; Week 12; Test type: Superiority; p = 0.0392, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = 1.59, 95% CI 2-sided [0.08 to 3.09]

20. Secondary Outcome: Change From Baseline in Female Sexual Function Index Domain Scores at Week 12
Description: The Female Sexual Function Index consists of 19 questions, organized into 6 domains (desire, arousal, lubrication, orgasm, satisfaction, and pain), answered by the participant on a scale from 1 to 5. Where relevant, some questions also include an option of 0 if not applicable due to no sexual activity. Each domain score was calculated by adding the scores of each item in the domain and multiplying by a domain factor. For all domains, higher values indicate better sexual function, according to the following:
  Desire (2 questions): domain score ranges from 1.2 to 6; Arousal (4 questions): domain score ranges from 0 to 6; Lubrication (4 questions): domain score ranges from 0 to 6; Orgasm (3 questions): domain score ranges from 0 to 6; Satisfaction (3 questions): domain score ranges from 0.8 to 6; Pain (3 questions): domain score ranges from 0 to 6.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available baseline and Week 12 data
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 303 | 308
units on a scale
  Desire: number analyzed (Participants) | 276 | 281
  Desire | 0.56 (0.07) | 0.39 (0.06)
  Arousal: number analyzed (Participants) | 276 | 280
  Arousal | 0.64 (0.11) | 0.44 (0.11)
  Lubrication: number analyzed (Participants) | 275 | 281
  Lubrication | 1.29 (0.12) | 0.89 (0.12)
  Orgasm: number analyzed (Participants) | 276 | 281
  Orgasm | 0.78 (0.12) | 0.63 (0.11)
  Satisfaction: number analyzed (Participants) | 262 | 271
  Satisfaction | 0.78 (0.09) | 0.62 (0.09)
  Pain: number analyzed (Participants) | 275 | 279
  Pain | 1.47 (0.12) | 1.01 (0.12)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Desire; Test type: Superiority; p = 0.0752, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = 0.16, 95% CI 2-sided [-0.02 to 0.34]
Statistical Analysis 2: Comparison: Ospemifene vs Placebo; Arousal; Test type: Superiority; p = 0.1867, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = 0.20, 95% CI 2-sided [-0.10 to 0.49]
Statistical Analysis 3: Comparison: Ospemifene vs Placebo; Lubrication; Test type: Superiority; p = 0.0161, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = 0.40, 95% CI 2-sided [0.07 to 0.73]
Statistical Analysis 4: Comparison: Ospemifene vs Placebo; Orgasm; Test type: Superiority; p = 0.3400, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = 0.16, 95% CI 2-sided [-0.16 to 0.48]
Statistical Analysis 5: Comparison: Ospemifene vs Placebo; Satisfaction; Test type: Superiority; p = 0.2195, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = 0.16, 95% CI 2-sided [-0.10 to 0.41]
Statistical Analysis 6: Comparison: Ospemifene vs Placebo; Pain; Test type: Superiority; p = 0.0103, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = 0.45, 95% CI 2-sided [0.11 to 0.80]

21. Secondary Outcome: Change From Baseline in Urinary Distress Inventory (UDI)-6 Total Score
Description: The presence or absence of urinary symptoms was assessed using the Urinary Distress Inventory (UDI)-6. The symptoms include frequent urination, urine leakage related to the feeling of urgency, urine leakage related to physical activity, coughing, or sneezing, small amounts of urine leakage, difficulty emptying bladder, and pain and discomfort in the lower abdominal or genital area. If a symptom was present, participants were asked to assess the degree to which they were bothered by it on the following 4-point scale:
  1. = present but doesn't bother her at all;
  2. = present and bothers her slightly;
  3. = present and bothers her moderately;
  4. = present and bothers her greatly. The total score was calculated by adding the 6 scores together (Absent = 0), and ranges from 0 to 24, with lower values indicating less urinary distress.
Time Frame: Baseline and Weeks 4, 8, and 12
Population: Intent-to-treat population with available data at each time point
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 311 | 314
units on a scale
  Week 4: number analyzed (Participants) | 295 | 298
  Week 4 | -0.8 (0.2) | -0.9 (0.2)
  Week 8: number analyzed (Participants) | 286 | 284
  Week 8 | -1.0 (0.2) | -1.4 (0.2)
  Week 12: number analyzed (Participants) | 275 | 280
  Week 12 | -1.3 (0.2) | -1.6 (0.2)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Week 4; Test type: Superiority; p = 0.7230, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = 0.1, 95% CI 2-sided [-0.4 to 0.6]
Statistical Analysis 2: Comparison: Ospemifene vs Placebo; Week 8; Test type: Superiority; p = 0.1104, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = 0.4, 95% CI 2-sided [-0.1 to 0.9]
Statistical Analysis 3: Comparison: Ospemifene vs Placebo; Week 12; Test type: Superiority; p = 0.2448, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = 0.3, 95% CI 2-sided [-0.2 to 0.9]

22. Secondary Outcome: Change From Baseline in Bone Sialoprotein at Week 12
Description: Serum bone sialoprotein (BSP) was measured as a marker of bone resorption.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available data
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 264 | 271
pg/mL | -24964.3 (3922.5) | -20576.1 (3871.5)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Test type: Superiority; p = 0.4263, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = -4388.3, 95% CI 2-sided [-15214.8 to 6438.3]

23. Secondary Outcome: Change From Baseline in Type I Collagen C-Telopeptide (CTX) at Week 12
Description: Type I collagen C-telopeptide was measured as a marker of bone resorption.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available data
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 261 | 260
ng/mL | -0.044 (0.008) | 0.006 (0.008)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = -0.049, 95% CI 2-sided [-0.071 to -0.027]

24. Secondary Outcome: Change From Baseline in Deoxypyridinoline at Week 12
Description: Deoxypyridinoline was measured as a marker of bone resorption.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available data
Measure: Least Squares Mean (Standard Error); unit: µmol/mol creatinine
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 261 | 260
µmol/mol creatinine | 0.08 (0.16) | 0.22 (0.16)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Test type: Superiority; p = 0.5159, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = -0.14, 95% CI 2-sided [-0.58 to 0.29]

25. Secondary Outcome: Change From Baseline in Type I Collagen N-Telopeptide (NTX) at Week 12
Description: Type I collagen N-telopeptide was measured as a marker of bone resorption.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available data
Measure: Least Squares Mean (Standard Error); unit: nmol bone collagen equivalents (BCE)/L
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 265 | 270
nmol bone collagen equivalents (BCE)/L | -0.10 (0.23) | 0.65 (0.23)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Test type: Superiority; p = 0.0227, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = -0.75, 95% CI 2-sided [-1.39 to -0.10]

26. Secondary Outcome: Change From Baseline in Tartrate-Resistant Acid Phosphatase 5b at Week 12
Description: Tartrate-resistant acid phosphatase 5b was measured as a marker of bone resorption.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available data
Measure: Least Squares Mean (Standard Error); unit: units/L
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 265 | 270
units/L | -0.28 (0.04) | -0.06 (0.04)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Test type: Superiority; p = 0.0003, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = -0.22, 95% CI 2-sided [-0.34 to -0.10]

27. Secondary Outcome: Change From Baseline in Alkaline Phosphatase at Week 12
Description: Alkaline phosphatase was measured as a marker of bone formation.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available data
Measure: Least Squares Mean (Standard Error); unit: units/L
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 258 | 261
units/L | -4.6 (0.7) | 1.6 (0.7)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = -6.2, 95% CI 2-sided [-8.1 to -4.3]

28. Secondary Outcome: Change From Baseline in Bone-specific Alkaline Phosphatase at Week 12
Description: Bone-specific alkaline phosphatase was measured as a marker of bone formation.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available data
Measure: Least Squares Mean (Standard Error); unit: units/L
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 265 | 270
units/L | -0.50 (0.36) | 0.84 (0.36)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Test type: Superiority; p = 0.0084, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = -1.35, 95% CI 2-sided [-2.35 to -0.35]

29. Secondary Outcome: Change From Baseline in Osteocalcin at Week 12
Description: Osteocalcin was measured as a marker for bone formation.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available data
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 265 | 270
ng/mL | -1.43 (0.31) | 0.62 (0.31)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = -2.06, 95% CI 2-sided [-2.92 to -1.19]

30. Secondary Outcome: Change From Baseline in Procollagen 1 N-Terminal Propeptide (P1NP) at Week 12
Description: Procollagen 1 N-terminal propeptide was measured as a marker of bone formation.
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available data
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 261 | 260
ng/mL | -3.22 (0.85) | 2.04 (0.86)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; The ANCOVA model included treatment group as a fixed effect and baseline value as a covariate; LS Mean Difference = -5.26, 95% CI 2-sided [-7.64 to -2.89]

31. Secondary Outcome: Mean Days of Lubricant Use Per Week
Description: The mean number of days/week that lubricant was used as documented by participants in an electronic daily diary.
Time Frame: Week 1 to Week 12
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 302 | 304
days/week | 0.8 (1.3) | 0.8 (1.2)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Test type: Superiority; p = 0.9575, Welch's t-test

32. Secondary Outcome: Mean Days of Intercourse Per Week
Description: The mean number of days/week of intercourse as recorded by participants in an electronic daily diary.
Time Frame: Week 1 to Week 12
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 302 | 304
days/week | 0.9 (1.0) | 0.9 (1.1)
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Test type: Superiority; p = 0.8772, Welch's t-test

33. Secondary Outcome: Overall Satisfaction With Treatment at Week 12
Description: Participants were asked to record their overall satisfaction with treatment in an electronic diary according to the following categories: Very satisfied, Moderately satisfied, About equally satisfied and dissatisfied, Moderately dissatisfied, and Very dissatisfied.
Time Frame: Week 12
Population: Intent-to-treat population with available data
Measure: Count of Participants; unit: Participants
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 221 | 198
Participants
  Very satisfied | 83 | 54
  Moderately satisfied | 71 | 52
  About equally satisfied and dissatisfied | 43 | 49
  Moderately dissatisfied | 13 | 26
  Very dissatisfied | 11 | 17
Statistical Analysis 1: Comparison: Ospemifene vs Placebo; Test type: Superiority; p = 0.0007, Wilcoxon rank-sum test

34. Secondary Outcome: Change From Baseline in Estradiol at Week 12
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 266 | 269
pg/mL | -2.5 (19.6) | 0.5 (10.3)

35. Secondary Outcome: Change From Baseline in Follicle-Stimulating Hormone at Week 12
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 268 | 270
IU/L | -5.18 (12.64) | -1.96 (11.79)

36. Secondary Outcome: Change From Baseline in Luteinizing Hormone at Week 12
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 266 | 270
IU/L | -1.58 (8.54) | -0.38 (7.59)

37. Secondary Outcome: Change From Baseline in Sex Hormone-Binding Globulin at Week 12
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 262 | 267
nmol/L | 30.44 (31.89) | 1.73 (17.61)

38. Secondary Outcome: Change From Baseline in Testosterone at Week 12
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 262 | 267
ng/dL | 1.1 (9.1) | 1.2 (20.2)

39. Secondary Outcome: Change From Baseline in Free Testosterone at Week 12
Time Frame: Baseline and Week 12
Population: Intent-to-treat population with available data
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Ospemifene | Placebo
Number analyzed (Participants) | 262 | 267
nmol/L | 0.0000 (0.0035) | 0.0007 (0.0115)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 14 days after the last dose; 14 weeks
Description: Participants who received at least 1 dose of study drug. Four participants randomized to placebo received ospemifene in error and are counted in the ospemifene group for safety assessments. One participant randomized to placebo who enrolled at 2 different sites at the same time was excluded.
Arm/Group | Ospemifene | Placebo
All-Cause Mortality (participants affected / at risk) | 0/317 | 0/310
Serious Adverse Events (participants affected / at risk) | 5/317 | 3/310
Other Adverse Events (participants affected / at risk) | 37/317 | 42/310
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ospemifene (N=317) | Placebo (N=310)
Bronchitis (Infections and infestations) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Transient global amnesia (Nervous system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ospemifene (N=317) | Placebo (N=310)
Nasopharyngitis (Infections and infestations) | 4 | 8
Upper respiratory tract infection (Infections and infestations) | 7 | 11
Urinary tract infection (Infections and infestations) | 7 | 10
Headache (Nervous system disorders) | 5 | 7
Hot flush (Vascular disorders) | 20 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-11-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT02638337/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT02638337/SAP_001.pdf